CLINICAL TRIAL: NCT02010398
Title: Neurophysiological, Dynamometric, Functional and Clinical Assessment of the Cross-Training Effect in Patients With Multiple Sclerosis
Brief Title: Effects of the Cross-Training in Patients With Multiple Sclerosis
Acronym: CTSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Professor Franca Deriu, Associate Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prot.1160/L
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis; Weakness; Fatigue
Keywords: Resistance training/methods; contralateral strength training; ipsilateral strength training; Isokinetic contraction; Adaptation, Physiological/physiology; Electromyography/methods; Transcranial Magnetic Stimulation/methods; Evoked Potentials, Motor
MeSH Terms: conditions — Multiple Sclerosis; Asthenia; Fatigue

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cross-Training healthy subjects (Active Comparator): A cohort of healthy subjects (N=15) will undergo a phase of intervention consisting of cross-training of the stronger limb employing an isokinetic contraction regimen at maximal intensity.
  Interventions: Other: Cross-Training healthy subjects
- Standard-Training multiple sclerosis (Active Comparator): A cohort of patients with multiple sclerosis (N=15), presenting with a marked asymmetry in limb strength, will undergo a standard-training of the more-impaired limb employing an isokinetic contraction regimen at maximal intensity.
  Interventions: Other: Standard-training multiple sclerosis
- Cross-Training multiple sclerosis (Experimental): A cohort of patients with multiple sclerosis (N=15), presenting with a marked asymmetry in limb strength, will undergo a cross-training of the less-impaired limb employing an isokinetic contraction regimen at maximal intensity.
  Interventions: Other: Cross-Training multiple sclerosis
- Healthy Control (No Intervention): A cohort of healthy subjects (N=15) will undergo baseline assessment and a second evaluation after one month of no-intervention

INTERVENTIONS:
Other: Cross-Training healthy subjects — The phase of intervention will consist of a 6-week cross-training of the stronger limb employing an isokinetic contraction regimen at maximal intensity.
  Arms: Cross-Training healthy subjects
Other: Cross-Training multiple sclerosis — The phase of intervention will consist of a 6-week cross-training of the less-impaired limb employing an isokinetic contraction regimen at maximal intensity.
  Arms: Cross-Training multiple sclerosis
Other: Standard-training multiple sclerosis — The phase of intervention will consist of a 6-week standard strength training of the more-impaired limb employing an isokinetic contraction regimen performed at maximal intensity.
  Arms: Standard-Training multiple sclerosis

SUMMARY:
The purpose of this study is to determine whether, in patients with multiple sclerosis presenting with marked asymmetry of strength, training the less-affected limb with a Cross-Training approach may induce a meaningful transfer of strength with neurophysiological, functional and clinical correlates, to the contralateral, more-impaired limb.

DETAILED DESCRIPTION:
Muscle weakness is a major disability that is responsible for deeply reducing the overall quality of life (QoL) of patients with Multiple Sclerosis (MS). Research has shown that strength training (ST) has a significant positive effect on the performance of daily living activities in people with MS, resulting in an increased QoL. Several ST methods are currently employed for reducing strength impairment in MS but no one regimen has been portrayed as superior to others. When strength impairment is prominently lateralized to one limb, training is commonly addressed to the weaker side in order to balance the deficit. However, such ST may not always be applicable to a severely weakened limb that is too compromised to sustain it. For these selected patients we hypothesize that training the less affected limb with a Cross Training (CT) approach may overcome the problem, also avoiding patients' frustration and potential withdrawals from rehabilitation programs.

Aim of this project is to investigate and compare in two groups of selected MS patients, with a marked asymmetry of strength, the effects induced on dynamometric, neurophysiological, functional and clinical outcomes by a CT of the less-impaired leg (CT group) compared to a ST of the more-impaired leg (ST group). In order to make comparisons with a population which is not exposed to the condition MS, a third group composed of healthy subjects will also be included in the study.

The research plan will be articulated in 5 phases (recruitment, baseline assessment, 6 week-intervention phase, post-intervention assessment and follow up at 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years
* Expanded Disability Status Scale (EDSS) ≤6 (Pyramidal functional system ≥3)

Exclusion Criteria:

* Clinically relevant cognitive disorders;
* Disability caused by other diseases;
* Medication with corticosteroids within three months prior to enrolment;
* Medication with botulinum toxin within six months prior to enrolment;
* Clinically or radiologically documented exacerbation within six months prior to enrolment;
* Variations in disease-modifying drugs (DMD) within three months prior to enrolment;
* Severe ataxia and postural instability (assessed with Berg Balance Scale);
* Depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-07; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Muscular strength | Muscular strength will be assessed at baseline, within one week from the completion of the 6-week rehabilitation phase and at 12-week follow up.
  Strength changes in the weaker side compared to the contralateral, through isokinetic dynamometry.

SECONDARY OUTCOMES:
Neural adaptations to Cross Training | Neural adaptations will be assessed at baseline, within one week from the completion of the 6-week rehabilitation phase and at 12-week follow up.
  Neural adaptations to CT occurring at cortical and/or spinal level, through transcranial magnetic stimulation (TMS) and peripheral electrophysiological recordings.

OTHER OUTCOMES:
Walking performance | It will be assessed at baseline, within one week from the completion of the 6-week rehabilitation phase and at 12-week follow up.
  Regarding the clinical and functional relevance to MS patients, changes from baseline in walking performance will be assessed through 6-Minute Walking Test (6MWT), which has been demonstrated to be a feasible, reproducible and reliable measure in MS and to be strongly correlated to subjective measures of ambulation; 10 Meter-Walk Test (10MWT), which estimates the walking speed at both comfortable and maximal velocities.
Fatigue | Assessment at baseline, within one week from the completion of the 6-week rehabilitation phase and at 12-week follow up.
  Modified Fatigue Impact Scale (MFIS): extracted from the Multiple Sclerosis Quality of Life Inventor. It consists of 21 items and provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning.
Executive functions | Assessment at baseline, within one week from the completion of the 6-week rehabilitation phase and at 12-week follow up.
  Frontal Assessment Battery (FAB): it tests executive functions, in a form of an interview with 6 functional tasks covering 5 domains: memory, planning, attention, reflex and visual spatial. The FAB correlates with dysfunction in a variety of cognitive domains including attention, memory, and executive functions.
Spasticity symptom severity | Assessment at baseline, within one week from the completion of the 6-week rehabilitation phase and at 12-week follow up.
  Modified Ashworth Scale: it is a widely used qualitative scale for the assessment of spasticity symptom severity and measures resistance to passive stretch, scoring from 0 (no increase in tone) to 4 (affected parts rigid in flexion or extension).
Gait Analysis for patients with Multiple Sclerosis | At baseline and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Franca Deriu, MD; PhD, Study Director — University of Sassari-Department of Biomedical Sciences
Locations (3):
- Italy (3):
  - Department of Biomedical Sciences- University of Sassari, Sassari, Sassari (SS)
  - Department of Clinical and Experimental Medicine, University of Sassari, Sassari
  - Department of Surgery, Microsurgery and Medical-Surgical Specialties, Sassari

REFERENCES:
- [Result] Manca A, Pisanu F, Ortu E, De Natale ER, Ginatempo F, Dragone D, Tolu E, Deriu F. A comprehensive assessment of the cross-training effect in ankle dorsiflexors of healthy subjects: A randomized controlled study. Gait Posture. 2015 Jun;42(1):1-6. doi: 10.1016/j.gaitpost.2015.04.005. Epub 2015 Apr 20. PMID 25922111
- [Derived] Morrone M, Martinez G, Achene A, Scaglione M, Masala S, Manca A, Deriu F. Size and site matter: the influence of corpus callosum subregional lesions on the magnitude of cross-education of strength. Front Physiol. 2025 Feb 24;16:1554742. doi: 10.3389/fphys.2025.1554742. eCollection 2025. PMID 40066282
- [Derived] Manca A, Martinez G, Aiello E, Ventura L, Deriu F. Effect of Eccentric Strength Training on Elbow Flexor Spasticity and Muscle Weakness in People With Multiple Sclerosis: Proof-of-Concept Single-System Case Series. Phys Ther. 2020 Jul 19;100(7):1142-1152. doi: 10.1093/ptj/pzaa055. PMID 32266379
- [Derived] Manca A, Martinez G, Cereatti A, Della Croce U, Ventura L, Dvir Z, Deriu F. Isokinetic predictors of gait speed increase following high-intensity resistance training of the ankle dorsiflexors in people with multiple sclerosis: A pilot study. Clin Biomech (Bristol). 2019 Jul;67:102-106. doi: 10.1016/j.clinbiomech.2019.05.008. Epub 2019 May 9. PMID 31100700
- [Derived] Manca A, Cabboi MP, Dragone D, Ginatempo F, Ortu E, De Natale ER, Mercante B, Mureddu G, Bua G, Deriu F. Resistance Training for Muscle Weakness in Multiple Sclerosis: Direct Versus Contralateral Approach in Individuals With Ankle Dorsiflexors' Disparity in Strength. Arch Phys Med Rehabil. 2017 Jul;98(7):1348-1356.e1. doi: 10.1016/j.apmr.2017.02.019. Epub 2017 Mar 23. PMID 28342828
- [Derived] Manca A, Dvir Z, Dragone D, Mureddu G, Bua G, Deriu F. Time course of strength adaptations following high-intensity resistance training in individuals with multiple sclerosis. Eur J Appl Physiol. 2017 Apr;117(4):731-743. doi: 10.1007/s00421-017-3534-z. Epub 2017 Mar 1. PMID 28251398
- [Derived] Manca A, Ginatempo F, Cabboi MP, Mercante B, Ortu E, Dragone D, De Natale ER, Dvir Z, Rothwell JC, Deriu F. No evidence of neural adaptations following chronic unilateral isometric training of the intrinsic muscles of the hand: a randomized controlled study. Eur J Appl Physiol. 2016 Oct;116(10):1993-2005. doi: 10.1007/s00421-016-3451-6. Epub 2016 Aug 2. PMID 27485469
- [Derived] Manca A, Cabboi MP, Ortu E, Ginatempo F, Dragone D, Zarbo IR, de Natale ER, Mureddu G, Bua G, Deriu F. Effect of Contralateral Strength Training on Muscle Weakness in People With Multiple Sclerosis: Proof-of-Concept Case Series. Phys Ther. 2016 Jun;96(6):828-38. doi: 10.2522/ptj.20150299. Epub 2015 Dec 4. PMID 26637645
- See also: A comprehensive assessment of the cross-training effect in ankle dorsiflexors of healthy subjects: A randomized controlled study. — https://www.ncbi.nlm.nih.gov/pubmed/25922111?report=docsum&format=text